CLINICAL TRIAL: NCT04886167
Title: A Dose-Ranging Study to Evaluate the Safety and Efficacy of AbobotulinumtoxinA for the Treatment of Moderate to Severe Platysmal Bands
Brief Title: Dysport Dose-Ranging Treatment of Platysmal Bands
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinical Testing of Beverly Hills (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CTBH-01-2021
Record Dates: First submitted 2021-05-05; First posted 2021-05-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Platysma Bands
Keywords: AbobotulinumtoxinA; Platysmal Bands
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 120U abobotulinumtoxinA (Active Comparator): Treatment of platysmal bands using a total of 120 U abobotulinumtoxinA. This will involve 24 injection sites (6 injections per each of 4 platysmal bands), with each injection site receiving 0.025mL (5 U).
  At the 14 day visit, an optional touch-up using up to 90 U of abobotulinumtoxinA can be performed. This will involve up to 18 injection sites, with each injection site receiving 0.025mL (5 U).
  Interventions: Drug: AbobotulinumtoxinA
- 180U abobotulinumtoxinA (Active Comparator): Treatment of platysmal bands using a total of 180 U abobotulinumtoxinA. This will involve 24 injection sites (6 injections per each of 4 platysmal bands), with each injection site receiving 0.0375mL (7.5 U).
  At the 14 day visit, an optional touch-up using up to 90 U of abobotulinumtoxinA can be performed. This will involve up to 12 injection sites, with each injection site receiving 0.0375mL (7.5 U).
  Interventions: Drug: AbobotulinumtoxinA
- 240U abobotulinumtoxinA (Active Comparator): Treatment of platysmal bands using a total of 240 U abobotulinumtoxinA. This will involve 24 injection sites (6 injections per each of 4 platysmal bands), with each injection site receiving 0.05mL (10 U).
  At the 14 day visit, an optional touch-up using up to 120 U of abobotulinumtoxinA can be performed. This will involve up to 12 injection sites, with each injection site receiving 0.05mL (10 U).
  Interventions: Drug: AbobotulinumtoxinA

INTERVENTIONS:
Drug: AbobotulinumtoxinA — Injection of platysmal bands.
  Other Names: Dysport

SUMMARY:
This is a double-blinded, dose-ranging study in the US to assess the efficacy, safety, and duration of response of abobotulinumtoxinA for the treatment of moderate to severe platysmal bands.

DETAILED DESCRIPTION:
This study is intended to evaluate the efficacy and safety of an initial dose of 120 U, 180 U, and 240 U of abobotulinumtoxinA (with optional touch-up) in the treatment of moderate to severe platysmal bands. The platysmal bands will be treated by intramuscular injection of abobotulinumtoxinA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 65 years of age.
2. Moderate to severe platysmal bands (grade 3 or 4 on the Photographic Platysma Bands Scale, which ranges from 1 [minimal] to 5 [extreme]) at rest and at maximum contraction as assessed by the Investigator Live Assessment (ILA).
3. Females of non-childbearing potential (i.e., post-menopausal [absence of menstrual bleeding for 1 year prior to screening, without any other medical reason], or has undergone hysterectomy or bilateral oophorectomy) or

   Females of childbearing potential with a negative urine pregnancy test at screening and baseline, and agrees to use a highly effective and approved contraceptive method for the duration of the study. A highly effective method of contraception is defined as:
   1. Bilateral tubal ligation;
   2. Combined (estrogen and progesterone containing) oral, intravaginal or transdermal contraceptives that inhibit ovulation as the primary mode of action, on a stable dose for at least 28 days prior to screening visit;
   3. Intrauterine device (IUD) inserted at least 28 days prior to screening visit;
   4. Intrauterine hormone-releasing system;
   5. Partner vasectomized for at least three months prior to screening visit;
   6. Progestogen -only oral, injectable or implantable contraceptives that inhibit ovulation as the primary mode of action, on a stable dose for at least 28 days prior to screening visit; or prior to screening visit; or
   7. Strict abstinence (i.e., refraining from heterosexual intercourse for the entire duration of the subject's participation in the study).
4. Time and ability to complete the study and comply with instructions.
5. Understands the study requirements and signed the informed consent form (ICF).

Exclusion Criteria:

1. Botulinum toxin treatment of any serotype below the lower orbital rim, in the neck or chest within 12 months prior to study treatment.
2. Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than the investigational product).
3. Known hypersensitivity to any component of the study product, or allergy to cow's milk protein* (according to the package insert/information).

   *This criterion does not exclude subjects who are lactose intolerant. Lactose intolerance is a gastrointestinal disorder caused by an enzyme deficiency (lactase). An allergy to cow's milk protein is an immunological disorder that results in a systemic reaction, such as anaphylaxis.
4. Known allergy or sensitivity to any botulinum toxin serotype.
5. Female who is breast-feeding.
6. Female who intends to conceive a child during the study.
7. Current smoker of any kind (e.g., tobacco, cloves, marijuana, vape pens, hookah, etc.), and agrees not to smoke for the duration of the study.
8. Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy to the lower face (i.e., below the level of the bottom of the nose), neck or chest within 12 months prior to study treatment.
9. Previous use of any permanent (non-biodegradable) or semi-permanent (e.g., calcium hydroxylapatite, Poly-L-lactic acid, polymethyl methacrylate, etc.) facial tissue augmentation therapy, lifting sutures, permanent implants or autologous fat to the lower face (i.e., below the level of the bottom of the nose), neck or chest within 24 months prior to study treatment.
10. History of lower face (i.e., below the level of the bottom of the nose), neck or chest surgery, aesthetic procedures (e.g. ablative skin resurfacing, laser, microneedling, chemical peel, micro-focused ultrasound, deoxycholic acid injections, micro-needling, non- surgical fat reduction procedure) in the previous 12 months, or any other procedures which the Investigator's opinion would interfere with study evaluations.
11. Planned surgery or aesthetic procedures to the lower face (i.e., below the level of the bottom of the nose), neck or chest (e.g. ablative skin resurfacing, laser, mesotherapy, Platelet-Rich Plasma (PRP) treatment, chemical peel, micro-focused ultrasound, deoxycholic acid injections, micro-needling, non-surgical fat reduction procedure) during the study period.
12. Clinically significant abnormal focused physical examination finding(s) at screening or baseline visits.
13. History of clavicular or sternal fracture.
14. Presence of inflammation, active infection or skin disorder, such as eczema, rosacea, psoriasis, pseudofolliculitis barbae, herpes zoster etc, near (i.e., superior to the clavicle and inferior to the mandible) or in the platysmal bands area.
15. History of neck pain, cervical disc degeneration, cervical dystonia, previous cervical neck surgeries, arm pain, numbness or weakness, asthenia, generalized muscle weakness, diplopia, blurred vision, ptosis, dysphagia, dysphonia, dysarthria, urinary incontinence, or breathing difficulties.
16. History or presence of cancerous or pre-cancerous lesions, or radiation near (i.e., superior to the clavicle and inferior to the mandible) or in the platysmal bands area.
17. Marked lower face (i.e., below the level of the bottom of the nose) or neck asymmetry, excessive neck skin or subcutaneous neck fat; excessive skin laxity, sagging, or banding; or deep horizontal neck folds.
18. Presence of scars, hair, or tattoos (facial, neck or chest) in the treatment area that may interfere with study evaluations.
19. History of bleeding disorder or current use of anticoagulant.
20. History or presence of any medical condition that may put the subject at increased risk with exposure to botulinum toxin including diagnosed myasthenia gravis, Lambert-Eaton- syndrome, amyotrophic lateral sclerosis, voice disorders (aphonia, dysphonia, etc.), stroke, facial nerve palsy, or any other condition that might interfere with neuromuscular function.
21. Use of medications that affect neuromuscular transmission such as curare-like depolarizing agents, lincosamides, polymyxins, anticholinesterases, and aminoglycoside antibiotics.
22. Use of a muscle relaxant within 2 weeks prior to study treatment or planned use during the study.
23. Treatment with any investigational drug or device within 30 days prior to study treatment.
24. Any prior or current psychiatric illness (e.g. psychosis, depression, anxiety), alcohol or drug abuse, or is taking antidepressant, anxiolytic, or antipsychotic medication that, in the Investigator's opinion, could affect the subject's safety and/or the conduct or outcome of the study.
25. Other concurrent medical conditions, therapy or other condition that, in the Investigator's opinion, would interfere with the evaluation of the study medication safety or efficacy and/or put the subject at risk if he/she participates to the study.
26. Study center personnel, close relatives of the study center personnel (e.g. parents, children, siblings, or spouse), employees or close relatives of employees at the Sponsor company.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Investigator Live Assessment (Dynamic) - 1 month | 1 month
  Responder rate at 1 month using the Investigator Live Assessment 5-point Photographic Scale at maximum contraction. The scale ranges from 1 to 5, with higher scores meaning a worse outcome.

SECONDARY OUTCOMES:
Investigator Live Assessment (Dynamic) | 5 months
  Responder rate at each post-treatment visit using the Investigator Live Assessment 5-point Photographic Scale at maximum contraction. The scale ranges from 1 to 5, with higher scores meaning a worse outcome.
Subject Self Assessment (Dynamic) | 5 months
  Responder rate at each post-treatment visit using the Subject Self Assessment 5-point Photographic Scale at maximum contraction. The scale ranges from 1 to 5, with higher scores meaning a worse outcome.
Investigator Live Assessment (At Rest) | 5 months
  Responder rate at each post-treatment visit using the Investigator Live Assessment 5-point Photographic Scale at rest. The scale ranges from 1 to 5, with higher scores meaning a worse outcome.
Subject Self Assessment (At Rest) | 5 months
  Responder rate at each post-treatment visit using the Subject Self Assessment 5-point Photographic Scale at rest. The scale ranges from 1 to 5, with higher scores meaning a worse outcome.
Response Duration | 5 months
  Time to loss of a grade 1 or 2 for both Investigator Live Assessment Scale and Subject Self Assessment Scale at maximum contraction and at rest. The scale ranges from 1 to 5, with higher scores meaning a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: John Joseph, MD, Principal Investigator — Principal Investigator
Locations (1):
- Clinical Testing of Beverly Hills, Encino, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monheit GD, Pickett A. AbobotulinumtoxinA: A 25-Year History. Aesthet Surg J. 2017 May 1;37(suppl_1):S4-S11. doi: 10.1093/asj/sjw284. PMID 28388718
- [Background] Carruthers J, Carruthers A. The evolution of botulinum neurotoxin type A for cosmetic applications. J Cosmet Laser Ther. 2007 Sep;9(3):186-92. doi: 10.1080/14764170701411470. PMID 17763029
- [Background] Matarasso A, Matarasso SL, Brandt FS, Bellman B. Botulinum A exotoxin for the management of platysma bands. Plast Reconstr Surg. 1999 Feb;103(2):645-52; discussion 653-5. doi: 10.1097/00006534-199902000-00043. PMID 9950556
- [Background] Brandt FS, Bellman B. Cosmetic use of botulinum A exotoxin for the aging neck. Dermatol Surg. 1998 Nov;24(11):1232-4. doi: 10.1111/j.1524-4725.1998.tb04103.x. PMID 9834744
- [Background] Kane MA. Nonsurgical treatment of platysmal bands with injection of botulinum toxin A. Plast Reconstr Surg. 1999 Feb;103(2):656-63; discussion 664-5. doi: 10.1097/00006534-199902000-00045. PMID 9950557